CLINICAL TRIAL: NCT00918099
Title: The Use of Avaulta for Anterior Repair. A Multicenter Randomised Prospective Controlled Study
Brief Title: The Use of Avaulta for Anterior Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Martin Rudnicki, ass. professor, Dept of Obstetrics and Gyneoclogy, Roskilde University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Avaulta
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Vaginal Prolapse
Keywords: Mesh; vaginal prolapse; Recurrence rate
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avaulta mesh (Active Comparator): Avaulta mesh
  Interventions: Procedure: Avaulta mesh
- Anterior repair (Active Comparator): Anterior repair
  Interventions: Procedure: Anterior repair

INTERVENTIONS:
Procedure: Avaulta mesh — Insertion of a mesh vs conventional repair
  Arms: Avaulta mesh
Procedure: Anterior repair — Conventional repair
  Arms: Anterior repair

SUMMARY:
Summary:

Vaginal prolapse is a well-known disease and is observed in approximately 11% of all postmenopausal women and tending to increase with age. Consequently, many surgical procedures have been developed in order to ensure sufficient support for the bladder, rectum or vaginal vault depending on the site of the defect. However, many procedures are associated with a high recurrence rate up to 40 % even within one to two years after the surgical procedure.

Due to the high recurrence rate new methods include the use of mesh, either biologically or synthetic. The latter is a permanent implant and therefore theoretically may result in a long-lasting anatomically correct position of the prolapse.

Although the recurrence rate may be lower using a mesh such surgical procedures may be associated with adverse events such as erosions of the vaginal mucosa. Others have observed shrinkage of the vaginal mucosa. However, in these studies large prolene mesh have been used. In contrast the recurrence rate is lowered up to 25%.

The above-mentioned advantage of synthetic mesh is however, mostly based on few non-randomised studies. The investigators therefore find it of importance to evaluate whether a surgical procedure using a mesh implant is superior to conventional surgical techniques. The present study is a clinical controlled study where patients with anterior vaginal prolapse are randomised to either a mesh technique or a standard anterior procedure.

The present study includes only two more visits at the outpatient clinic after the surgical procedure. Furthermore the patients have to fulfil questionnaires regarding urinary and faecal leakage and sexual habits.

Any participation in the study is totally voluntary and the patient may at any time withdraw herself. In any case the patient will receive the investigators' standard treatment.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL:

The use of Avaulta for anterior repair. A multicenter randomised prospective controlled study.

BACKGROUND:

During the resent years the methods for pelvic organ prolapse repair have changed rapidly. The reason for this is several. Firstly, there is a relative high recurrence rate in patients having an anterior vaginal repair. Thus, the rate has been estimated to be close to 40% or even higher and most often the recurrences occurs within the first two years. Weber et al and Sand et al reported various techniques of the anterior colporrhaphy without the use of mesh to be successful in the management of cystoceles in only 42 and 57%, respectively. In contrast others have shown a much lower 1-year recurrence rate. Shull reported on the safety and efficacy of the paravaginal repair but this procedure may also vary in success from 67 - 100%. Taken all together however, interpretation of these studies is difficult since the patients included have undergone at least one (in most cases several) vaginal surgical procedures at the same time and some studies even include patients with recurrence together with patients scheduled for primary vaginal surgery. Secondly, there is a need for simple procedures, which can be performed in an outpatient clinic and thirdly, the surgery should be acceptable for the women, i.e. without postoperative pain, short recovery period and no need for further surgical intervention.

In most centers a vaginal surgical repair of an anterior genital prolapse is performed in a standard manner through a midline incision followed by dissection of the vaginal mucosa from the pubocervical fascia. Interrupted sutures approximating the fascia at the midline then repair the cystocele. However, this may not be sufficient in those cases where no fascia is present or the presence of huge defects in the pubocervical fascia. As a consequence the use of mesh have been more popular. Several studies report a reduced recurrence rate following anterior repair using different types of mesh such as biomesh (6,7) or nonabsorbable mesh. The latter has been shown to be associated with vaginal erosion 8 - 2%%, which probably is related to the strong inflammatory response observed after implementation of such mesh. Another complication is shrinkage of the vaginal mucosa and this may be followed by sexual dysfunction or dyspareunia.

Polypropylene mesh appears to induce less inflammatory respons compared to other types. A specific type of mesh is the Avaulta Biosynthetic Mesh, which is a polypropylene mesh coated with collagen. This layer protects against inflammatory response and is slowly resolved.

Since most studies have included patients undergoing several vaginal surgical procedures at the same time, it is difficult to conclude whether or not the use of mesh is superior compared to conventional technique. Furthermore, only sparse information is available regarding sexual function and dyspareunia following vaginal prolapse surgery. Especially there is a lack of information regarding new mesh types.

The purpose of the present study is therefore to test the hypothesis that the Avaulta Biosynthetic Mesh is associated with a lower recurrence rate after two years of follow-up compared to conventional anterior repair. Secondly, the study is planned to evaluate the frequency of sexual dysfunction following vaginal anterior repair, and if there is any difference between the two surgical methods.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 55 yr
* Women with anterior vaginal wall prolapse stage >2 according to POP-Q classification
* Good understanding the language in word and writing

Exclusion Criteria:

* A history of pervious major pelvic surgery with the exception of a hysterectomy for reasons other than genital prolapse
* Patients with previous vaginal surgery because of defects in the anterior of posterior compartments
* Previous hysterectomy because of vaginal prolapse
* Patients with prolapse of uterus or an enterocele > stage 1
* Patients with previous TVT performed through the obturator membrane
* History of genital or abdominal cancer
* Patients treated with corticostaroids
* Not able to understand the study protocol (language problems, cognitive dysfunction etc.)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Does Avaulta reduce the recurrence rate | 0ct 2008 - July 2010

SECONDARY OUTCOMES:
Does Avaulta improve prolapse symptoms, quality of life and sexual function | oct 2008-July 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Roskilde University Hospital, Roskilde, Denmark